CLINICAL TRIAL: NCT00004336
Title: Pilot Study of Familial Nonsyndromal Mondini Dysplasia
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Other Study IDs: 199/11895; UMMC-1402
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Mondini Dysplasia
Keywords: Mondini dysplasia; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Genetic Diseases, Inborn; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Determine the mode of inheritance of nonsyndromal Mondini inner ear dysplasia, an inner ear malformation causing deafness, vestibular dysfunction, and recurrent meningitis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

The parents of 1 family with known Mondini dysplasia are screened for the disorder using temporal bone computerized tomography without contrast. This information is used to determine the mode of inheritance.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Parents of a study family with nonsyndromal Mondini dysplasia

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2
Dates: Start 1995-10

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Griffith, Study Chair — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States